CLINICAL TRIAL: NCT05053828
Title: Impact of Type 2 Diabetes on Outcomes Associated With Antiplatelet Drugs: A Retrospective Analysis
Brief Title: Type 2 Diabetes With Antiplatelet Drugs
Status: Completed | Type: Observational
Sponsor: Tabula Rasa HealthCare (Industry)
Responsible Party: Sponsor
Other Study IDs: TRHC-T2D-2021-001
Record Dates: First submitted 2021-09-13; First posted 2021-09-23 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Type2 Diabetes; Antiplatelet Drugs; Myocardial Infarction; Heart Failure
MeSH Terms: conditions — Myocardial Infarction; Heart Failure | interventions — Platelet Aggregation Inhibitors; Clopidogrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-diabetic controls on clopidogrel: Non-diabetic patients prescribed clopidogrel
  Interventions: Drug: Antiplatelet Drug
- Diabetic patients on clopidogrel: Diabetic patients on clopidogrel
  Interventions: Drug: Antiplatelet Drug
- Diabetic patients on antiplatelet drugs other than clopidogrel: Diabetic patients on antiplatelet drugs other than clopidogrel
  Interventions: Drug: Antiplatelet Drug

INTERVENTIONS:
Drug: Antiplatelet Drug — Antiplatelet drugs and agents
  Other Names: Clopidogrel

SUMMARY:
Tabula Rasa HealthCare (TRHC), d/b/a CareKinesis, is the first national pharmacy that provides science-based medication risk identification and mitigation technologies and services. CareKinesis utilizes medication decision support tools and pharmacists certified in geriatrics to provide pharmacy services for various healthcare organizations including PACE organizations (described above). Presently, CareKinesis services more than 35 PACE organizations, including approximately 140 PACE sites, across the country. As a national PACE pharmacy provider since 2011, CareKinesis focuses on improving medication regimens to reduce medication-related risks while enhancing economic, clinical and humanistic outcomes. Pharmacist-led clinical services and medication safety reviews are currently being offered to PACE organizations under the direction of licensed healthcare prescribers by TRHC (CareKinesis). Through mutual data-sharing agreements, patient data will be collected retrospectively for patients satisfying the inclusion and exclusion criteria.

TRHC via other programs such as the Center for Medicare & Medicaid Enhanced Medication Therapy Management program with BlueCross BlueShield Northern Plain Alliance and ClearStone, or via collaboration as third party with other health plans can have access to de-identified patient's data. TRHC has also established an agreement with the Watson IBM database to retrieve relevant patients' information for research.

DETAILED DESCRIPTION:
This research is a retrospective observational study which does not involve interaction neither intervention with any subjects or their treatment. Using deidentified data, we plan to collect information about every subject including but not limited to demographic information (age, gender, race), drug claims, health outcomes and disease outcomes (using ICD10 codes), and cost. Data will be collected from the time patient enrolled in PACE in partnership with TRHC or from other health care plans working in collaboration with TRHC. Subjects prescribed antiplatelet agents will be identified. ICD10 codes will be used to determine disease conditions (type 2 diabetes, type 1 diabetes, non-diabetic). Next, patients prescribed clopidogrel will be identified from patients prescribed alternate anti-platelet therapy (excluding aspirin). For each cohort, Major Adverse Cardiac Event (MACE) outcomes, hospitalization data relating to bleeding incidents, stent thrombosis, mortality due to cardiovascular events, and all-cause mortality outcomes will be extracted from ICD10 codes and health insurance data. Using the medication list, the medication risk score (MRS®) and cost data will be extracted and analyses will be conducted to address our study objectives.

ELIGIBILITY:
Inclusion Criteria:

* Patient is enrolled in a healthcare organization where TRHC provides pharmacy services during the implementation period; or patient's data enrolled with health plan organization having partnership with TRHC; or patient's data from the IBM Watson database.
* Patient must be taking anti-platelet medication including clopidogrel, prasugrel, and ticagrelor during the period in which data is collected.

Exclusion Criteria:

* Patients not taking above mentioned anti-platelet medications during the period in which data is collected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PACE population is adults aged 55 years and older who are eligible for Medicare and Medicaid.
Sampling Method: Probability Sample
Enrollment: 173464 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Measure the prevalence of clopidogrel prescription in patients with T2D in the study population. | 1 year
  Quantitative
Measure the prevalence of ticagrelor and prasugrel prescription in patients with T2D vs. clopidogrel. | 1 year
  Quantitative
Calculate MedWise Risk Score (TM) of <10, 11-14, 15-19, 20-30, >30 for T2D patients to examine patient risk for adverse drug events. | 1 year
  Quatitative

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Michaud, Principal Investigator — Tabula Rasa HealthCare
Locations (1):
- Tabula Rasa Healthcare, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No